CLINICAL TRIAL: NCT06423300
Title: Evaluation of the Patellar LIFT System for Subjects With Patellofemoral Cartilage Degeneration
Acronym: PELICAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZKR Orthopedics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP0001
Record Dates: First submitted 2024-04-24; First posted 2024-05-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group: LIFT (Experimental): Subjects receiving the LIFT implant system.
  Interventions: Device: LIFT Implant
- Control Group: TTO (Active Comparator): Subjects receiving a Tibial Tubercle Osteotomy (TTO)
  Interventions: Other: Tibial Tubercle Osteotomy

INTERVENTIONS:
Device: LIFT Implant — The LIFT implant provides a less invasive option for treatment of patellofemoral cartilage degeneration in the knee. the LIFT implant unloads the patellofemoral joint by elevating the patellar tendon to unload the joint compartment and realign the kneecap toward healthier cartilage
  Arms: Treatment Group: LIFT
Other: Tibial Tubercle Osteotomy — Tibial Tubercle Osteotomy
  Arms: Control Group: TTO

SUMMARY:
The PELICAN study is a prospective, non randomized, dual arm, multi-center clinical study comparing clinical outcomes of subjects treated with the LIFT Implant System to subjects treated with Tibial Tubercle Osteotomy (TTO).

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 22 to 65 years at time of screening
2. Anterior knee pain due to patellofemoral cartilage degeneration (PCD) with an Modified Outerbridge score of ≥3 as assessed by an MRI on the study knee
3. Body Mass Index (BMI) of ≤ 35
4. Weight < 300 lbs
5. Anterior Knee Pain Score (AKPS) of ≤ 70 (0-100 scale)
6. Visual Analog Score (VAS) of ≥ 40 (0-100 scale)
7. Failure of at least 6 months of non-surgical treatment defined as at least one of the treatments (e.g. rest, bracing, physical therapy, targeted exercise, use of NSAIDs, activity level reduction or Confidential ZKR Orthopedics, CIP 0001 Page 11 of 55 Protocol Version: 1.0, 04JAN2024 modification, etc.) per AAOS Treatment of Osteoarthritis of the Knee; Evidence based guideline 3rd Edition 2021

Exclusion Criteria:

1. PCD with an Modified Outerbridge Score of 2 or less at the study knee
2. Clinical symptoms of the contralateral knee that preclude activities of daily living, stair climbing, stair descending, or require the use of an assist device
3. History of patella dislocation or instability
4. Patella alta or patella baja
5. Known TT-TG distance >20mm
6. Patients requiring simultaneous cartilage grafting procedure, cartilage transplantation, or bone marrow stimulation
7. Previous repair of a torn patellar tendon
8. Prior TTO procedure or knee joint replacement (total or partial) of the study knee
9. Joint modifying surgery (e.g., ligament reconstruction, meniscus repair, cartilage transplantation, microfracture, etc.) in the study knee within 6 months prior to planned index procedure date
10. Arthroscopic surgeries in the study knee for joint lavage, meniscectomy, chondral debridement, and loose body removal within 3 months prior to planned index procedure
11. Active infection, sepsis, osteomyelitis or history of septic arthritis in any joint
12. Rheumatoid arthritis, other forms of inflammatory joint disease or autoimmune disorder
13. History of avascular necrosis of any bone
14. History of symptomatic patellar tendonitis of intrasubstance tear
15. Insufficiency of the cruciate, collateral ligaments, or tendon which would preclude stability of the LIFT System
16. Pathologic ligamentous injury (Lachman > 1) or meniscus tearing
17. Clinical symptoms of the femoral-tibial joint of the study knee that preclude activities of daily living, stair climbing, stair descending, or requires the use of an assist device
18. Evidence (MRI, arthroscopy, etc.) of Modified Outerbridge Grade 4 degenerative arthritis in the femoral-tibial joint of the study knee that potentially explains patient symptoms

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
24 month composite endpoint demonstrating non-inferiority of the LIFT System as compared to TTO. | 24 months
  The Composite Endpoint is comprised of the following:
  1. an improvement of >10 points from baseline in the Anterior Knee Pain Scale (AKPS)
  2. Freedom from serious procedure-related adverse events leading to secondary surgical intervention (SSI).
  3. As determined by x-ray or MRI: Freedom from loosening of implant, loosening of bone screws, breakage of screw or implant, migration of implant; TTO osseous non-union, partial union, delayed union, malunion in any plane, TTO screw loosening, TTO screw breakage
  The above 3 measures are COMBINED to produce the composite endpoint. If the subject meets all 3 outcome measures above at the 24 month mark - the outcome is listed as "non inferiority of the LIFT System as compared to TTO"

SECONDARY OUTCOMES:
Time to Partial Weight Bearing (Recovery) | 24 months
  Superiority of the LIFT system to TTO data for the length of time it takes for a subject to return to partial weight bearing.
Time to Full Weight Bearing Without Assistive Devices (Recovery) | 24 months
  Superiority of the LIFT system to TTO data for the length of time it takes for a subject to return to full weight bearing without the use of assistive devices.
Function | 3 Months
  Superiority of the LIFT system to TTO data for:
  Functional Outcome: Early Functional Improvement as determined by the baseline change of the AKPS (Anterior Knee Pain Scale) Score. The AKPS is graded on a scale of 0 to 100, with 100 being the highest possible score.
Function | 24 Months
  Superiority of the LIFT system to TTO data for:
  Functional Outcome: Late Functional Improvement as determined by the baseline change of the AKPS Score (Anterior Knee Pain Scale) Score. The AKPS is graded on a scale of 0 to 100, with 100 being the highest possible score.
Patient's Reported Pain Level | 3 Months
  Superiority of the LIFT system to TTO data for:
  Early pain improvement as determined by a 30% or more improvement from baseline in knee pain score at 3 months
Patient's Reported Pain Level | 24 Months
  Superiority of the LIFT system to TTO data for:
  Late pain improvement as determined by a 30% or more improvement from baseline in knee pain score at 24 months

OTHER OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 months
  Patient Report Outcome KOOS Survery
Level of Patient Satisfaction (Patient Reported) | 24 months
  This outcome will determine the patient's satisfaction with the procedure based on a patient reported satisfaction questionnaire.
Willingness of Patient to Have Procedure Again (Patient Reported) | 24 months
  This outcome will determine the patient's willingness to repeat the LIFT procedure based on a patient reported questionnaire.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Horizon Clinical Research, La Mesa, California
  - Hospital for Special Surgery, New York, New York
  - NYU Langone Health, New York, New York
  - Ohio State University - Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No